CLINICAL TRIAL: NCT02522130
Title: Different Analgesics Prior to IUD Insertion: Is There Any Evidence?
Brief Title: Different Analgesics Prior to Intrauterine Device (IUD) Insertion: Is There Any Evidence?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Hayat National Hospital (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, mohamed maher, assistant professor, Al Hayat National Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ob/gyn4
Record Dates: First submitted 2015-07-08; First posted 2015-08-13 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: IUD Insertion Complication
MeSH Terms: interventions — Lidocaine; Misoprostol; Naproxen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- lidocaine group (Active Comparator): Group A will receive 10 ml 1% lidocaine (Xylocaine 1%, Astra Zeneca, Egypt) Para cervical block prior to insertion of IUD (injection sites at cervix-vaginal junction typically at 4 ,8 O'clock), Then 3 minutes waiting period between the administration of the Para cervical block and IUD insertion,
  Interventions: Drug: Lidocaine
- misoprostol group (Active Comparator): Group B will receive 400 mcg oral misoprostol (Sigma, Egypt) prior to IUD insertion
  Interventions: Drug: oral misoprostol
- non steroid group (Active Comparator): Group C will receive oral naproxen (Naprosyn, Syntax, Egypt) prior to IUD insertion
  Interventions: Drug: naproxen
- placebo group (Placebo Comparator): group D will receive placebo tablets.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Lidocaine — intracervical injection
  Arms: lidocaine group
Drug: oral misoprostol — oral treatment
  Arms: misoprostol group
Drug: naproxen — oral treatment
  Arms: non steroid group
Other: placebo — oral treatment
  Arms: placebo group

SUMMARY:
Different ways of reducing pain during IUD insertion have been explored. So a randomized study will be conducted to test their role

DETAILED DESCRIPTION:
A randomized clinical controlled trial of women undergoing IUD insertion. Participants in the study groups will be randomly assigned by labeled opaque envelopes to either1% lidocaine (Xylocaine 1%, Astra Zeneca, Egypt), misoprostol (Sigma, Egypt), naproxen (Naprosyn, Syntax, Egypt) or placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

Patients are considered eligible if:

1. they are alert oriented and co-operative to response to the visual analogue scale (VAS).
2. They will sign the informed consent to participate in the clinical trial before entering the study.
3. Willingness to be randomized and complete study questionnaires.

Exclusion Criteria:

Participants are excluded from participation if they are ineligible for an IUD by accepted criteria of our institution such as:

1. A lidocaine allergy
2. Copper allergy
3. Current cervicitis
4. Pelvic inflammatory disease (PID) within 3 months
5. Uterine anomalies
6. Pain medication within 6 hours before insertion
7. Misoprostol administration within 24 hour before insertion
8. History of cervical surgery and contraindication to study medications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
current pain level with IUD insertion and 15 minutes post procedure measured by the Visual Analogue Scale. | 15 minutes
  A Visual Analogue Scale is a measurement instrument that tries to measure a characteristic or attitude that is believed to range to across a continuum of values and can not easily to be directly measured. Subjects pain using a 10 point visual analogue scale (-+VAS, anchors: 0=non, 10 = worst imaginable).
  The participants were asked to mark their pre IUD insertion pain expectancies initially, then to mark their pain during different steps of IUD placement.

CONTACTS AND LOCATIONS:
Locations (2):
- Menoufia University, Shebin Elkom, Egypt
- Alhayah national hospital, Abhā, Saudi Arabia